CLINICAL TRIAL: NCT05510297
Title: Development of a Comprehensive, Active Seating System to Lessen Sedentariness and Improve Health and Wellness in Older Adults: In-home Testing Phase
Brief Title: Active Seating System to Lessen Sedentariness in Older Adults: In-home Testing Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stacey L. Schepens Niemiec, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP-22-00037; R43AG074697 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-home feasibility test (Other): In this single-arm trial, participants will use an active seating system for a 3- to 7-day period. The system provides a seating platform and treadles to pedal while in a seated or semi-reclined position. The system will also include a digital user interface to track performance.
  Interventions: Device: FitSitt Prototype

INTERVENTIONS:
Device: FitSitt Prototype — FitSitt merges features of a posture chair, exercise machine, and tracking means. It provides seated stepping, postural support, and semi-recline capabilities. A digital interface and app will allow users to set goals and track performance.

SUMMARY:
FitSitt is an innovative device tailored to older adults that increases the convenience of breaking up sedentary activity and incorporating physical activity into in-home daily routines. This comprehensive seating solution merges features of a posture chair, exercise machine, rehabilitation tool, and activity tracker. Its primary purpose is to reduce daily immobile time, offering users a convenient means for replacing sedentary bouts with varying intensities of physical activity, ultimately leading to improved health. FitSitt aims to improve the baseline activity profile of its users by providing a comprehensive wellness solution including a non-disruptive in-home means for physical activity engagement while allowing users to continue participation in desired seated activities. In so doing, FitSitt has the potential to decrease health-harmful sedentary activity in a wide variety of high-risk individuals and occupational contexts. The initial development of FitSitt for this Phase I proposal, however, will target community-dwelling older adults.

Co-led by Activ Sitting, Inc. and USC, Phase I will include three study phases (i.e., focus group, in-lab testing, in-home testing) to determine user acceptability, feasibility of procedures, safety, and preliminary efficacy to affect health and behavior outcomes. Clinical trial activities occur within the in-home testing stage and will focus on user acceptability and preliminary efficacy to affect health and behavioral outcomes. This information will be used along with other information collected from the overall study to redesign and enhance the current FitSitt prototype and prepare the system to be tested in a fully powered Phase II study of the enhanced FitSitt's efficacy to improve health in community-living older people. As currently designed, FitSitt provides convenience, comfort, and health value-add for myriad older adults, ensuring scalability and sustainability of broad use across communities and markets. This project will facilitate the development of an optimized, in-home, comprehensive sedentary activity solution for older adults and countless other populations that could benefit from reducing the deleterious health effects of extended inactive behavior through convenient and comfortable-to-use intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years old or older
2. English-speaking
3. Live in local Los Angeles area and no plans to vacation away from home during the trial period
4. Self-reported ability to safely engage in 30 minutes of light-intensity activity per day
5. Self-reported ability to pedal comfortably without stopping for 5 minutes
6. Community-dwelling

Exclusion Criteria:

1. Dependence in transferring to a chair safely
2. Inability to safely and reliably access and operate FitSitt (ascertained by a brief demonstration at beginning of in-home visit)
3. A member living in the same household participated in the in-home testing stage of this study
4. Participated in the in-lab testing stage of the study already
5. Unstable health conditions such as uncontrolled blood pressure, end-stage renal failure on renal replacement therapy, or malignancy currently on chemotherapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Schepens Niemiec, PhD, Principal Investigator — University of Southern California Chan Division of OS-OT
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
This proposal will produce proprietary data relevant to the patented FitSitt system owned by Activ Sitting, Inc. Under the Small Business Act, SBIR/STTR grantees are protected from disclosure and nongovernmental use of all SBIR/STTR data developed from work performed under a SBIR funding agreement for a period of 20 years after the closeout of a Phase I trial. Accordingly, the team will not engage in data sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 screened for enrollment; 12 screen failures; 17 enrolled by signing consent and beginning at least one baseline survey activity; 15 began the intervention period (2 had withdrawn prior to the intervention beginning).
Period: Overall Study
Arm/Group | In-home Feasibility Test
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [70 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 7
  Race/ethnicity: Non-Hispanic Black | 2
  Race/ethnicity: Latino/Hispanic | 2
  Race/ethnicity: Asian | 4
Region of Enrollment [Number; unit: participants]
  United States | 15
Daily hours reported watching TV [Median (Inter-Quartile Range); unit: Hours/day] | 3 [2 to 5]
Confidence using a smartphone [Median (Inter-Quartile Range); unit: units on a scale] — Self-reported confidence in using a smartphone generally on a scale of 1=poor to 10=excellent.
  units on a scale | 7 [6 to 8]
Smartphone operating system [Count of Participants; unit: Participants] — Population: Not all participants reported having a smartphone; smartphone ownership was not a requirement of the study.
  Participants
    number analyzed (Participants) | 11
    Android | 3
    iOS | 8
Years of smartphone ownership [Median (Inter-Quartile Range); unit: years] — Population: Not all participants owned a smartphone; this was not a requirement for the study. Only those who owned a smartphone were reported here.
  years
    number analyzed (Participants) | 11
    (all) | 13 [8 to 18]
Health conditions [Number; unit: participants] — Only health conditions that were self-reported by 3 or more participants are listed here.
  participants
    Arthritis | 9
    High cholesterol | 5
    Osteoporosis / osteopenia | 5
    High blood pressure | 5
    Cancer | 4
    Diabetes (I or II) | 3

OUTCOME MEASURES:

1. Primary Outcome: Daily Prolonged Sedentary Bouts (activPAL+FitSitt Sensors) Change From Baseline to up to 7 Days With Intervention Present
Description: Daily prolonged sedentary bouts (objective sedentary activity) will be measured in real time using the activPAL thigh-worn accelerometer during a 72-hour monitoring period before introduction of FitSitt (i.e., pre-intervention) and throughout a 3- to 7-day long monitoring period when FitSitt is present (i.e., intervention-present). "Prolonged" sedentary bouts is identified by an activPAL proprietary algorithm of sedentariness >= 30 minutes in duration, and will be merged with data captured with FitSitt sensors when sitting in the FitSitt. Bouts will be expressed in hours per 24-hour period.
Time Frame: Intervention-present monitoring period (3-7days) relative to pre-intervention 72-hour baseline
Measure: Median (Inter-Quartile Range); unit: hours/24-hr period
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 13
hours/24-hr period | -1.7100 [-3.1700 to -0.4450]
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney); Median Difference (Net) = 7.000

2. Secondary Outcome: Daily Steps Change From Baseline to up to 7 Days With Intervention Present
Description: Daily Steps (objective physical activity) will be measured in real time using the activPAL thigh-worn accelerometer during a 72-hour monitoring period pre-intervention and throughout a 3- to 7-day long monitoring period when the intervention is present. "Steps" (i.e., pedaling counts) accumulated while sitting and using FitSitt will be merged with the activPAL data. Daily steps are expressed in counts per 24-hour period.
Time Frame: Intervention-present monitoring period (3-7days) relative to pre-intervention 72-hour baseline
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 14
steps per day | 3142.88 (5277.55)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.074, t-test, 2 sided — a priori threshold for statistical significance=0.05 for 2-sided t-test; no adjustments for multiple comparisons made; data were checked for normality using the Shapiro-Wilk test where p>0.05 was interpreted as likely normal distribution; Mean Difference (Final Values) = 2653.16, 95% CI 2-sided [-297.76522 to 5604.07522], Standard Deviation 5110.86

3. Secondary Outcome: Self-reported Physical Activity Change From Baseline to 3-7 Days
Description: Self-reported physical activity will be measured via the Physical Activity Scale for the Elderly (PASE). PASE is a ten-item instrument designed to assess engagement in physical activities commonly pursued by older adults, including those related to leisure, household, and occupational tasks. The tool is a valid and reliable measure of physical activity engagement in the older adult population. Scores range from 0 to 361. Higher scores indicate a higher level of activity.
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | 4.44 (41.59)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority — a priori threshold for statistical significance=0.05 for 2-sided t-test; no adjustments for multiple comparisons made;; p = 0.685, t-test, 2 sided; Mean Difference (Net) = 4.44067, 95% CI 2-sided [-18.59116 to 27.47249], Standard Deviation 41.59009

4. Secondary Outcome: Self-reported Fatigue Severity Change From Baseline to 3-7 Days
Description: Fatigue will be measured using the Brief Fatigue Inventory, a 9-item questionnaire that captures subjective report of fatigue severity. It takes approximately 5 minutes to complete. This tool demonstrates good psychometric properties and is sensitive to change. Higher scores indicate greater fatigue. Scores range from 0 to 10 (mean of 9 items on a 0-10 scale).
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | -0.51 (1.45)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.191, t-test, 2 sided; Mean Difference (Net) = -0.51267, 95% CI 2-sided [-1.31374 to 0.28841], Standard Deviation 1.44656

5. Secondary Outcome: Self-reported Pain Severity Change From Baseline to 3-7 Days
Description: Pain severity will be assessed using two Brief Pain Inventory (BPI) - Short Form subscales: severity. The severity subscale measures amount of pain presently and at its "worst," "least," and "average" severity. This subscale is considered valid and reliable. Higher scores = greater pain severity. Scores range from 0 to 10 and are calculated using the mean of the items.
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | -0.45 (1.35)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.218, t-test, 2 sided; Mean Difference (Net) = -0.45000, 95% CI 2-sided [-1.19775 to 0.29775], Standard Deviation 1.35026

6. Secondary Outcome: Self-reported Pain Interference Change From Baseline to 3-7 Days
Description: Pain interference will be assessed using the Brief Pain Inventory (BPI) - Short Form subscale: pain interference. The interference subscale assesses how much a person's pain disrupts everyday life. This subscale is considered valid and reliable. Higher scores indicate greater pain interference. Scores range from 0 to 10 and are calculated using the mean of the items.
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | -0.92 (2.19)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.125, t-test, 2 sided; Mean Difference (Net) = -0.92400, 95% CI 2-sided [-2.13898 to 0.29098], Standard Deviation 2.19396

7. Secondary Outcome: Self-reported Joint Stiffness Change From Baseline to 3-7 Days
Description: The Musculoskeletal Stiffness Questionnaire (MSQ) is a 21-item patient-reported outcome measure that takes approximately ≤10 minutes to complete. It assesses joint stiffness and the physical and psychosocial impact of stiffness on daily life. Items are scored on a Likert scale, and the raw scores are transformed into a total percentage score ranging from 0 to 100, with higher scores indicating greater joint stiffness and worse outcomes. Validation studies have included healthy adults across the lifespan as well as persons with rheumatoid arthritis and chikungunya disease. The total score is derived by summing item responses, converting the total to a percentage of the maximum possible score. If subscale scores are reported, each subscale score also ranges from 0 to 100.
  Unit of Measure: Scores on a scale from 0-100
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
percent | 0.0013 (0.10148)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.960, t-test, 2 sided; Mean Difference (Net) = 0.00133, 95% CI 2-sided [-0.05486 to 0.5753], Standard Deviation 0.10148

8. Secondary Outcome: FitSitt Seat Occupancy Usage Behavior
Description: FitSitt seat occupancy usage behavior is defined as number of minutes spent sitting in FitSitt across a 24-hour day, as captured by onboard FitSitt sensors. Users will have FitSitt available to them for 3 to 7 days.
Time Frame: From baseline through 3-7 days (daily)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
minutes per day | 214.20 (139.22)

9. Secondary Outcome: FitSitt Pedaling Usage Behavior
Description: FitSitt pedaling usage behavior is defined as number of minutes spent pedaling while seated in FitSitt across a 24-hour day, as captured by onboard FitSitt sensors. Users will have FitSitt available to them for 3 to 7 days.
Time Frame: From baseline through 3-7 days (daily)
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 14
minutes per day | 101.3 (65.95)

10. Secondary Outcome: FitSitt Use Self-efficacy
Description: FitSitt use self-efficacy will be assessed using a study-specific adaptation of the Self-Efficacy for Exercise scale, which we have entitled FitSitt Use Self-efficacy. Items have been modified to focus on using FitSitt as the mode of sedentary activity disruption rather than addressing exercise in general terms. The form is expected to take approximately 3 minutes to complete. Higher scores would indicate greater self-efficacy to use the device. Scores range from 0 to 10 and are calculated using the mean of the items.
Time Frame: 3-7 days (post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | 7.66 (2.58)

11. Secondary Outcome: Fatigue Interference Change
Description: as for outcome 4
Time Frame: Baseline and 3-7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-home Feasibility Test
Number analyzed (Participants) | 15
score on a scale | -0.51 (1.45)
Statistical Analysis 1: Comparison: In-home Feasibility Test; Test type: Superiority; p = 0.168, t-test, 2 sided; Mean Difference (Net) = -0.62200, 95% CI 2-sided [-1.53867 to 0.29467], Standard Deviation 1.65530

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | In-home Feasibility Test
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-home Feasibility Test (N=17)
Skin irritation activPAL (Skin and subcutaneous tissue disorders) | 1 (1) — Participant reported skin irritation and warmth from the activPAL activity monitor to the thigh.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT05510297/Prot_SAP_002.pdf
  • Informed Consent Form (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05510297/ICF_001.pdf